CLINICAL TRIAL: NCT06667492
Title: Reliability and Validity of Lower Extremity Dynamometry Assessment in Neurotypical Children
Brief Title: Lower Extremity Dynamometry Assessment in Neurotypical Children
Status: Recruiting | Type: Observational
Sponsor: University of Thessaly (Other)
Responsible Party: Principal Investigator, George Paras, Assistant Professor, University of Thessaly
Other Study IDs: dynam-neurotyp-child
Record Dates: First submitted 2024-10-27; First posted 2024-10-31 (Actual); Last update posted 2025-12-29 (Actual); Status verified 2025-12

CONDITIONS: Force Measurement; Children; Lower Limb; Assessment Tool
Keywords: dynamometry; lower limb; assessment; child

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Neuro-typical Children: Typically developing children aged 5 to 16 years with the ability of voluntary motor control are in included in the study.
  Interventions: Device: Traction Dynamometry

INTERVENTIONS:
Device: Traction Dynamometry — K-Pull dynamometer (Model MP.09.02.FN, Kinvent, Montpellier, France) is an assessment tool used to quantify muscle strength. It uses traction through a non-elastic strap to facilitate isometric contractions. This instrument will be used to evaluate isometric activity (maximum and average torque values) of the hip and knee flexors and extensors at specific joint angles.

SUMMARY:
The purpose of this study is to assess the reliability (intra-rater and inter-rater) and criterion validity (using a Cybex isokinetic dynamometer as the reference) of the K-Pull (traction) dynamometer for evaluating lower limb function in children with neurotypical development.

ELIGIBILITY:
Inclusion Criteria:

* typically developing children,
* between the ages of 5 and 16 years,
* have the capacity for voluntary motor control

Exclusion Criteria :

* undergone any treatment or intervention that could impact neuromuscular performance, such as surgery or medication use,
* experienced a recent injury
* demonstrating low levels of compliance during assessments are not included in the study.

Ages: 5 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: The study population consists of typically developing children aged 5 to 16 years, selected based on specific inclusion and exclusion criteria to ensure the reliability and validity of traction dynamometry.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2024-09-20 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Average Peak Torque | Through study completion, an average of 5 months
  Average Peak Torque refers to the average highest force output recorded during isometric contractions and represents the maximal strength generated by the muscle group being assessed (e.g., hip or knee flexors and extensors). Unit of Measure: Newton-metre (Nm)

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Physiotherapy - University of Thessaly, Lamia, Phthiotis, Greece

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hebert LJ, Maltais DB, Lepage C, Saulnier J, Crete M. Hand-Held Dynamometry Isometric Torque Reference Values for Children and Adolescents. Pediatr Phys Ther. 2015 Winter;27(4):414-23. doi: 10.1097/PEP.0000000000000179. PMID 26397089
- [Background] Daloia LMT, Leonardi-Figueiredo MM, Martinez EZ, Mattiello-Sverzut AC. Isometric muscle strength in children and adolescents using Handheld dynamometry: reliability and normative data for the Brazilian population. Braz J Phys Ther. 2018 Nov-Dec;22(6):474-483. doi: 10.1016/j.bjpt.2018.04.006. Epub 2018 May 4. PMID 29802034